CLINICAL TRIAL: NCT00586014
Title: High Dose Sequential Therapy and Autologous Stem Cell Rescue for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0074
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Autologous Stem Cell Transplant
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): High-dose sequential cyclophosphamide and VP-16 followed by myeloablation with high-dose BCNU and melphalan with autologous stem cell transplant
  Interventions: Procedure: High-Dose Sequential Chemotherapy followed by ASCT

INTERVENTIONS:
Procedure: High-Dose Sequential Chemotherapy followed by ASCT — Patient will receive Cyclophosphamide(4 g/m2 over 2 hours) and blood progenitor cell collection (day -49). G-CSF (10 mcg/kg/d) will be administered SQ. A six hour leukapheresis will be performed,cells will undergo CD34+ cell selection, patients will receive high dose VP-16 (Etopophos)(day -28)(2 g/m2 over 4 hours)and G-CSF (5 mcg/kg/d) will be administered SQ two days following VP-16. The an IV of sulfamethoxazole-trimethoprim 1 ampule BID for 5 days (Day -5). BCNU 500 mg/m2 IV over 2 hours (Day -4). Melphalan (Day -2) will be administered IV (200 mg/m2 over 20 minutes). The frozen peripheral blood mononuclear cells will be transfused on Day 0. Day +1: G-CSF 5 mcg/kg/d SQ for 3 days.

SUMMARY:
The purpose of this phase II study is to assess the toxicity and efficacy of sequentially administered high dose chemotherapy followed by autologous stem cell rescue in the treatment of multiple myeloma. Prior studies have shown that dose-intensified melphalan can produce higher response rates and complete remission in some patients. Over the past several years, multiple phase II studies utilizing high dose chemotherapy or high dose chemo-radiotherapy with autologous marrow or peripheral blood stem cell rescue have demonstrated improved response rates and survival rates compared to historical controls. Recently a prospective randomized trial has demonstrated improved response rates, response duration and overall survival utilizing high dose therapy with autologous bone marrow support compared to standard chemotherapy. The primary cause of failure is relapse and it is unclear how many, if any, patients are cured by this approach. Based on observations of efficacy in Hodgkin's Disease, Non-Hodgkin's Lymphoma, and breast cancer, an approach utilizing sequential high dose chemotherapy in multiple myeloma was developed. This protocol tests the sequential regimen in multiple myeloma patients who have responded to a standard dose chemotherapy regimen prior to enrollment.

DETAILED DESCRIPTION:
The purpose of this phase II study is to assess the toxicity and efficacy of sequentially administered high dose chemotherapy followed by autologous stem cell rescue in the treatment of multiple myeloma. Multiple myeloma is a chemotherapy sensitive disease but is not curative with standard therapy with a median survival of 2 to 4 years. Prior studies have shown that dose-intensified melphalan can produce higher response rates and complete remission in some patients. Over the past several years, multiple phase II studies utilizing high dose chemotherapy or high dose chemo-radiotherapy with autologous marrow or peripheral blood stem cell rescue have demonstrated improved response rates and survival rates compared to historical controls. Recently a prospective randomized trial has demonstrated improved response rates, response duration and overall survival utilizing high dose therapy with autologous bone marrow support compared to standard chemotherapy. The primary cause of failure is relapse and it is unclear how many, if any, patients are cured by this approach. Based on observations of efficacy in Hodgkin's Disease, Non-Hodgkin's Lymphoma, and breast cancer, an approach utilizing sequential high dose chemotherapy in multiple myeloma was developed. This protocol tests the sequential regimen in multiple myeloma patients who have responded to a standard dose chemotherapy regimen prior to enrollment. As originally written, eligible patients were required to have sensitive disease.

The protocol was revised in August 1998 to allow entry of patients with newly diagnosed myeloma who had stable but not progressive disease following VAD chemotherapy. Patients with recurrent myeloma were still required to have chemotherapy sensitive disease. Eligible patients must also have pathologically confirmed multiple myeloma, no prior bone marrow transplantation and acceptable organ function (pulmonary, renal, hepatic, and cardiac). The recent revision of the protocol also allows entry of patients with renal insufficiency due to multiple myeloma to be enrolled on the protocol. Prior to initiating high dose therapy, patients must undergo a complete history and physical exam with routine lab work plus titers for HIV, CMV, HSV, and VCV: immunoglobulin levels, beta-2 microglobulin and serum protein electrophoresis as well as immunoelectrophoresis and bone marrow aspirates and biopsies. These studies are all standard for multiple myeloma patients. All patients require a double Human Hickman to be placed prior to the start of therapy. The protocol was originally written to include total body irradiation and high dose Melphalan as a preparative regimen for patients who had not received prior radiotherapy. Patients who were not eligible for TBI received high dose BCNU plus Melphalan. A revision removed the TBI Melphalan arm from the protocol after analysis of over 100 patients treated at Stanford University Medical Center on this same protocol showed no difference in event-free survival or overall survival between the TBI containing arm and the chemotherapy only preparative regimen. The TBI arm was dropped due to the increased cost and morbidity of TBI and the associated scheduling and logistics problems. The other revision to the protocol was the inclusion of CD34 stem cell selection on the stem cells collected by leukapheresis following high dose cyclophosphamide. This change was based on the results of a Phase III study which demonstrated that the degree of tumor cell contamination of these stem cell collections could be decreased by 3-6 logs with CD34 cell selection. The dose of Melphalan was also increased to 200 mg/m2 after completion of a dose escalation study at Stanford.

ELIGIBILITY:
Inclusion Criteria:

* All patients must receive multi-agent based chemotherapy, preferably VAD, as cytoreduction prior to transplantation. The time from the last chemotherapy administration must be greater than 21 days. Patients with recurrent myeloma must have sensitive disease as demonstrated by a decrease in serum or urine paraprotein levels of >50% or a decrease in bone marrow plasmacytosis to less than 20%. Patients with newly diagnosed myeloma may have stable (but not progressive) disease following VAD.
* Patients must have their pathology reviewed and the diagnosis of multiple myeloma confirmed at the transplant center. Patients with smoldering multiple myeloma or benign monoclonal gammopathy of unknown significance will be excluded from this study.
* Performance status: -CALGB 0.1 or Karnofsky greater than 70%
* Patients must have serum creatinine < 2 x upper limit of normal, bilirubin < 2 x upper limit of normal, transaminases < 2 x upper limit of normal, MUGA resting EF > 50% or more than a 5% increase with exercise if <50%, DLCO > 60%

Exclusion Criteria:

* Patients who have undergone bone marrow transplantation previously will not be eligible.
* Patients with HIV, HBsAG positive
* Pregnant or lactating women
* Patients with other medical or psychiatric disorders which would seriously compromise tolerance to this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 1997-05; Primary Completion 2006-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the progression free survival at one year in multiple myeloma patients who receive sequentially administered high dose cyclophosphamide and VP-16 followed by high-dose BCNU (Carmustine) plus Melphalan | 4 years

SECONDARY OUTCOMES:
To evaluate the response rates of multiple myeloma patients to this sequentially administered high dose chemotherapy. | 4 years
To evaluate the safety and toxicity of this sequential high dose chemotherapy program in multiple myeloma patients. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Chao, MD, Principal Investigator — Duke Health